CLINICAL TRIAL: NCT05486819
Title: Effect of Lignocaine Versus Sodium Bicarbonate on Reducing Pain Due to Intravenous Injection of Propofol : a Prospective Randomised Double-blinded, Controlled Study
Brief Title: Lignocaine Versus Sodium Bicarbonate on Reducing Pain During Propofol Injection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Hussein, lecturer of anesthesia , surgical icu and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pain during propofol injection
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Propofol Adverse Reaction
Keywords: lignocaine,sodium bicarbonate,pain on propofol injection
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (L) (Active Comparator): receive 3 ml (60 mg) of lignocaine 2% added to propofol during injection
  Interventions: Drug: Propofol Injection
- Group (B) (Active Comparator): receive 3 ml of sodium bicarbonate 8.5% added to propofol during injection
  Interventions: Drug: Propofol Injection
- Group (S) (Placebo Comparator): receive 3 ml of normal saline added to propofol during injection
  Interventions: Drug: Propofol Injection

INTERVENTIONS:
Drug: Propofol Injection — adding lignocaine or sodium bicarbonate to propofol to reduce pain during injection

SUMMARY:
To compare the effect of adding lignocaine and sodium bicarbonate to propofol in reducing pain on propofol injection (POPI).

DETAILED DESCRIPTION:
Propofol is the most commonly used intravenous (IV) anesthetic drug for induction of anesthesia and for sedation. It is almost an ideal IV anesthetic agent, but pain which occur during its injection still remains a problem. This pain may not be a serious complication, but most patients remember it as an unpleasant encounter with anesthetists. In one survey, pain on propofol injection (POPI) stands 7th most important problem in the current practice of anesthesia . About 70 to 90% of patients who were given propofol for anesthesia induction experience pain during injection and this pain can be quite severe. All phenols irritate skin and mucous membranes. Thus, propofol being an alkyl-phenol is expected to induce pain despite the fact that it is almost isotonic. POPI has also been described as angialgia which means that the pain is due to vascular involvement . POPI is immediate as well as delayed after 10-20 seconds . The immediate pain is due to irritation of vein endothelium while as delayed pain is due to the release of mediators such a kininogen from kinin cascade . The most frequently used drug to alleviate POPI is intravenous lignocaine. The use of lignocaine to decrease POPI is due to its local anesthetic effect on the veins. However, it does not alleviate pain effectively in about 40% of the patients treated in this way (2). Administration of sodium bicarbonate was proved to reduce POPI. The proposed mechanism is through increasing sodium ions concentration as well as increasing serum pH through its buffering effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years old.
* Patients classified as ASA I or II.

Exclusion Criteria:

* Patients with the history of allergy to propofol or lignocaine.
* Patients took any medication for analgesia or sedation in the past 24 hours.
* Body mass index (BMI) more than 30.
* Patients classified as ASA III & IV.
* Severe mental illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
measuring the pain intensity immediately after intravenous injection of propofol using the four point verbal rating | 5 months

SECONDARY OUTCOMES:
1. Pain intensity at any top up doses of propofol. 2. Heart rate: baseline, 5 seconds, 1 minute & 5 minutes after injection. 3. Blood pressure: baseline, immediately after assessing the pain score then 5 minutes later | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No